CLINICAL TRIAL: NCT05199844
Title: Accuracy of Apple Watch to Measure Cardiovascular Indices in Patients With Cardiac Diseases: Observational Study
Brief Title: Smart Watch, Heart Rate and So2 in Cardiac Patients
Status: Completed | Type: Observational
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Alaa Khushhal, Principal Investigator, Umm Al-Qura University
Other Study IDs: HAPO-02-K-012
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Apple Watch
Keywords: Cardiac rehabilitation; Validity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group A: cardiac patients with regular heart rate
  Interventions: Device: Apple Watch
- Group B: cardiac patients with irregular heart rate

INTERVENTIONS:
Device: Apple Watch — Apple Watch device measures heart rate and oxygen saturation
  Groups: Group A

SUMMARY:
Background: Apple Watch validity to measure the heart rate (HR) and oxygen saturation (Spo2) in healthy subjects has been investigated, but its accuracy and validity for patients with cardiac diseases is still unclear. The HR is an important measure to determine the recommended exercise training intensity and to monitor the training intensity in patients with cardiac diseases. The target exercise training intensity during cardiac rehabilitation is between 40% to 70% of heart rate reserve (HRR). Also, cardiac patients who have hypoxemia are advised to continuously monitor their Spo2. Therefore, this study aims to investigate the accuracy of the Apple Watch in measuring the HR and Spo2 in Saudi patients with cardiac diseases.

Method: A cross sectional study will be invited one-hundred cardiac patients will be invited and recruited to participate in this study and the eligible participants will be randomly allocated into two groups. The first group (Group-A) will include the cardiac patients with regular HR and the second group (Group-B) will include the cardiac patients with irregular HR. Both groups will use the apple watch to evaluate the HR and the Spo2 against the Polar HR monitor and pulse oximeter at rest, during, and after the mild to moderate intensity exercise training session (40% to 70% HRR). The HR and the Spo2 monitoring, and recording will run on a 30 second schedule at rest (pre-session; for 3-minutes), during the 15-minutes session and over 5-minutes after the session). The main outcomes will be the HR and the Spo2 and will be evaluated before, during and after the exercise session using the Apple watch and the Polar HR monitor. All participants will receive the mild to moderate exercise training session (40 to 70 % HRR) using cycling and treadmill instruments for 15 minutes, proceeded, and followed by a 3-minutes warm-up and cool-down.

DETAILED DESCRIPTION:
Introduction:

Measuring the heart rate (HR) is important to estimate the suitable exercise training intensity and to determine the recommended exercise intensity (1). The 12-leads electrocardiogram (ECG) is the gold standers to measure heart rate, but it may be not suitable to be used outside the laboratory, therefore using the polar chest strap is the alternative to be used outside the lab and it has been tested against the 12-leads ECG during exercise and at rest in healthy subjects [2,3,4] and cardiac patients [5]. The HR following exercise is called heart rate recovery and it is important to predict mortality risk and cardiorespiratory fitness [6].

There is a liner relationship between the HR and oxygen consumption [7]. The Oxygen saturation (Spo2) is recommended to be monitored in patients with hypoxemia to extend their survival [8]. Some cardiac patients have hypoxemia particularly cardiac patients after cardiac arrest [9]. Pulse oximeter is a gold standard to measure the Spo2 [10].

The Apple Watch all versions can measure heart rate, but the latest versions-6 and 7 can measure blood Spo2. Photoplethysmography (PPT) is a non-invasive measurement procedure to evaluate the HR through wrist-worn devise by detecting each heartbeat changes in blood flow and changes colors in blood flow. The PPT has been used to measure Spo2, cardiac output, and blood pressure in many medical devices [11]. The PPT technology can help in early detection of some cardiovascular diseases such as atherosclerosis and atrial fibrillation [12].

A pilot study measured the HR agonist the telemetry in 50 cardiac patients (half of them with atrial fibrillation (AF) and other half with normal HR rhythm) during rest, through assessments of the HR 3-times/ day for two days. They found that the HR accuracy in patients with AF (r=86) was more than the cardiac patients who have normal rhythm (r= 0.64) and the overall accuracy was (r=070) but this still pilot study and more studies with large sample size are needed to confirm this findings in addition to presence of some limitations in this pilot study, as including of 3 black participants that could affect the accuracy of the results, presence of other interfering devices near the Apple Watches devices during evaluations in the cardiac wards and the fluid and edema after operation[13]. Moreover, the accuracy of the Apple Watch in measuring the HR during exercise is still unknown with cardiac patients and cardiac patients with AF.

Another study measured the HR from the Apple Watch against the 12-lead ECG during the cycle ergometer test for 30 seconds at three times (at rest (ICC=0.72), moderate exercise intensity (ICC=0.82), high exercise intensity (ICC=0.95)). The results revealed that the accuracy of Apple Watch has been increased with increasing exercise intensity in 40-patients with cardiovascular diseases, with good correlation at all three times [14].

A recent study measured the HR in 80 cardiac patients including some AF in phase-II or III in cardiac rehabilitation (exercises including steady cycle and treadmill). The study measured the HR from the limbs leads of ECG against the Polar HR, Apple Watch, Fitbit Blaze, Garmine Forerunner 235, and TomTom Spark Cardio (one instrument on each wrist), which means only 40-patients tested with the Apple Watch. They recorded the HR at rest and at 3, 5 and 7 minutes of cycle and Treadmill training. They found that the polar chest strap (r=0.99) was the most accurate during all exercises to the ECG followed by the Apple Watch (r=.80) and the Apple Watch accuracy during cycle increased to (r=0.89)[5]. However, the proportion of the AF in 80-patients was low (12 AF) and they were mix with the normal HR, so it could not know if the AF affect the accuracy of the Apple Watch or not and the 8-time points measured in this study was good, but if the study measured the heart rate every 15 or 10-seconds the results could be more meaningful. This study suggested that validation of the Apple Watch with AF should be investigated.

The new feature of measuring the blood Spo2 established in the Apple Watch is includes only on series 6 and 7. There is only one study examined the validity of the Apple Watch against two pulse oximeters to measure the Spo2 in 100-participants including 16-healthy subjects and 84-patients with medically controlled pulmonary diseases (including 23 patients with chronic obstructive pulmonary disease (COPD) and 61-patients with interstitial lung diseases. They found that the Apple Watch has strong positive correlations with the pulse oximeter (r=0.81, P<0.0001) [15]. Moreover, the study suggested to test the validity of the Apple Watch for measuring the blood Spo2 in other groups of patients.

The Apple Watch is a smart watch measuring the HR and the Spo2 but its validity in cardiac patients including patients with abnormal HR patterns is still unknown. Therefore, this will be the first study to evaluate the Apple Watch accuracy and validity for measuring the HR at rest, during and after exercises and to measure the Spo2 at rest and after exercises in patients with cardiac diseases including cardiac patients with normal HR and cardiac patients with abnormal HR patterns.

Method:

A cross sectional study will be invited one-hundred cardiac patients to participate in this study. The first group will be around 50 cardiac patients with sinus heart rhythm and the second group will be around 50 cardiac patients those with irregular heart rate. The distribution of patients into two groups will be based on the availability of the cardiac patients at Umm Al-Qura University Medical Center. Each participant will wear the Polar chest strap HR and the Apple Watch at rest, during exercises for 15 minutes and after exercises. The pulse oximeter will be used at rest and after exercises. The exercise session will be about 15-minutes duration at mild to moderate intensity according to the heart rate reserve (HRR) using the treadmill and the cycle ergometer, preceded by a 3-minutes warm-up, and followed by 3-minutes cool-down. The HR will be recorded every 30 seconds during whole period and the oxygen saturation will be recorded five times at rest and after exercises.

This study will follow the Declaration of Helsinki 1975 principles, revised in 2000 and will be conducted at the Umm Al-Qura University Medical Center, and will be in line with the Faculty of Applied Medical Sciences, Umm Al-Qura University ethical guidelines. Each participant will sign a written consent approving the volunteer participation in this study and agreeing for publication of its results. Suitable sample size was computed using the online G-power tool (https://download.cnet.com/G-Power/3000-2054_4-10647044.html), considering the effect size = 0.4, giving a sample size of 54 participants to provide reliable results. Extra-number will be included to substitute any participant's withdrawal or discontinuation.

Inclusion criteria: eligible participants will be cardiac patients as those with myocardial infarction (6-weeks post-insult), coronary bypass graft surgery (CABG), cardiac patients with valve diseases, stable atrial fibrillation (AF), heart failure (HF)-I,II and III, with and resting ejection fraction (EF) greater than 50%.

Exclusion criteria: Cardiac patients with unstable angina, uncontrolled high blood pressure, unstable arrhythmia, presence of complex ventricular arrhythmias, ST-segment depression ≥2mm from baseline during exercise testing or recovery, pacemaker patients will be all excluded from the study.

Risk management:

All measurements in this study will be done as the normal measurements for each cardiac patients who visited the Umm Al-Qura University Medical Center, so there is no risk for the patients to take part in this study. Moreover, the exercise intensity will determine for each patient, so each patient will do the exercise intensity that suitable for them. In case any terribly ill happen because of the study procedure, the cardiologist (Dr.Mahmoud) will be supervised each patients in this study.

Note: This study will not use any questionnaire to collect the data.

Data analysis:

All data will enter into the SPSS program for analyses. The results of this study may will analyze using the Pearson correlation test to test the difference between the Apple Watch and Polar heart rate for measuring heart rate and between the Apple Watch and Pulse oximeter for measuring SpO2 to test the validity. The P value will be set at 0.05 for significant results.

ELIGIBILITY:
Inclusion Criteria:

* eligible participants will be cardiac patients as those with myocardial infarction (6-weeks post-insult), coronary bypass graft surgery (CABG), cardiac patients with valve diseases, stable atrial fibrillation (AF), heart failure (HF)-I,II and III, with and resting ejection fraction (EF) greater than 50%.

Exclusion Criteria:

* Cardiac patients with unstable angina, uncontrolled high blood pressure, unstable arrythmia, presence of complex ventricular arrhythmias, ST-segment depression ≥2mm from baseline during exercise testing or recovery, pacemaker patients will be all excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac patients with sinus heart rate and irregular heart rate
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate | over 31 minutes
  Heart rate

SECONDARY OUTCOMES:
Spo2 | over 10 minutes at rest and after exercise
  Oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Umm Al-Qura University Medical Center, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The data may be published in research article or conference